CLINICAL TRIAL: NCT02600754
Title: Telehealth Treatments for Depression With Low-Income Homebound Seniors
Brief Title: Telehealth Depression Treatments for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Baylor College of Medicine (Other); University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Namkee Choi, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MD009675 (NIH)
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Depression
Keywords: older adults, depressive symptoms, psychosocial treatment
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IT-PST (Experimental): IT-PST refers to problem-solving therapy that will be tele-delivered by licensed mental health clinicians co-located in an aging-service agency (Meals on Wheels and More).
  Interventions: Behavioral: IT-PST
- IT-SCM (Experimental): IT-SCM refers to self-care management support that will be tele-delivered by trained lay advisers (TLAs) co-located in an aging-service agency (Meals on Wheels and More).
  Interventions: Behavioral: IT-SCM
- Wait-list control (Usual Care or UC) (No Intervention): Participants who will serve as controls with telephone safety calls

INTERVENTIONS:
Behavioral: IT-PST — 5 sessions of problem-solving therapy by licensed mental health clinicians co-located in an aging-service agency (Meals on Wheels and More)
  Arms: IT-PST
Behavioral: IT-SCM — 5 sessions of self-care management support by trained lay advisers co-located in an aging-service agency (Meals on Wheels and More)
  Arms: IT-SCM

SUMMARY:
This study aims to find an effective and sustainable approach to reducing disparities in accessing mental health services for an underserved and growing population group of low-income, racially diverse, homebound older adults. It will compare two aging-service integrated, teledelivered depression treatments for these seniors. One model is short-term problem-solving therapy by licensed clinicians; the second model is self-care management support by trained lay advisors. The findings are expected to create a foundation of information for guiding the implementation of acceptable, effective, and sustainable depression care within widely available aging-service infrastructures.

DETAILED DESCRIPTION:
The long-term objective of the proposed study is to improve access to depression treatments for low-income, racially diverse homebound seniors, a population experiencing significant disparities in mental health care due to their homebound and low-income status. Specific aims are to compare the acceptability, clinical effectiveness, treatment cost, and budget impact of the two teledelivered treatment delivery models: problem-solving therapy (PST) by licensed clinicians and self-care management (SCM) support by trained lay mental health workers/advisors. The interventionists will be integrated into an aging-service agency; hence, integrated tele-PST (IT-PST) ad integrated tele-SCM (IT-SCM). Although tele-psychotherapy is likely to be an effective mental health service delivery model for the target population, the current and projected shortage of such clinicians and the costs of deploying highly trained professionals pose barriers to this model's widespread real-world adoption and sustainability. A more plausible option may indeed have to utilize trained lay mental health workers. The study participants will be 276 low-income, racially diverse homebound seniors who are served by a home-delivered meal (HDM) program and other aging-service agencies in Austin, Tex. In a 3-arm, pragmatic clinical trial with randomization prior to consent (a preferred public health approach), the participants will receive five sessions of IT-PST, five sessions of IT-SCM, or five telephone check-in calls (for the usual care-UC-group). Our first hypothesis is that IT-PST and IT-SCM will be equally acceptable to the participants. Our second hypothesis is that both IT-PST and IT-SCM will be more effective than UC in reducing depressive symptoms, although IT-PST may be more effective than IT-SCM. Symptoms will be assessed with the 24-item Hamilton Depression Rating Scale (HAMD) at 12, 24, and 36 weeks after baseline. Additional outcomes will be depression-free days (DFDs) and disability (WHODAS 2.0). Our third hypothesis is that IT-SCM will have a lower delivery cost than IT-PST, but both IT-PST and IT-SCM will be more cost-effective than usual care. The analyses include (a) comparisons of delivery costs between IT-PST and IT-SCM; (b) assessment of cost-effectiveness (CEA) based on DFDs and health-related quality adjusted life-year measured by EuroQol-5 (EQ-5D); and (3) budget impact (BIA) of IT-PST relative to IT-SCM. Both CEA and BIA will employ a hybrid public program perspective of the AoA and the Centers for Medicare and Medicaid. Public health significance of this study is that the data will help aging-service providers and funders assess respective strengths and weaknesses of each model as a sustainable approach to providing depression care for an underserved and growing population group and improving their access to evidence-based mental health services. (The terms older adults and seniors are used interchangeably because the latter term is frequently used in aging services.)

ELIGIBILITY:
Inclusion Criteria:

* (1) HAMD >14; (2) age > 49; (3) English or Spanish Speaking; and (4) Non-Hispanic White, Black, or Hispanic

Exclusion Criteria:

* (1) antidepressant intake < 9 weeks; (2) high suicide risk; (3) probable dementia;( 4) bipolar disorder; and (5) substance use

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | 36 weeks
  24-item depression scale

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule | 36 weeks
  12-item disability assessment
Euro-Quol | 36 weeks
  measure of depression free days
Cornell Service Index | 36 week
  measure of physical and mental health, and social service use

CONTACTS AND LOCATIONS:
Overall Officials: Namkee G Choi, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Chen GJ, Kunik ME, Marti CN, Choi NG. Cost-effectiveness of Tele-delivered behavioral activation by Lay counselors for homebound older adults with depression. BMC Psychiatry. 2022 Oct 17;22(1):648. doi: 10.1186/s12888-022-04272-9. PMID 36253766
- [Derived] Choi NG, Marti CN, Wilson NL, Chen GJ, Sirrianni L, Hegel MT, Bruce ML, Kunik ME. Effect of Telehealth Treatment by Lay Counselors vs by Clinicians on Depressive Symptoms Among Older Adults Who Are Homebound: A Randomized Clinical Trial. JAMA Netw Open. 2020 Aug 3;3(8):e2015648. doi: 10.1001/jamanetworkopen.2020.15648. PMID 32865577